CLINICAL TRIAL: NCT00160576
Title: A Therapeutic Exploratory, Single Arm, Multicenter Trial to Evaluate the Efficacy and Safety of Levetiracetam up to 4000 mg/Day (500mg Oral Tablets) on Levodopa Induced Dyskinesias in Adults With Idiopathic Parkinson's Disease
Brief Title: Levetiracetam Treatment in Adult Subjects With Parkinson's Disease Experiencing Troublesome Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: N01105
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2009-09

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Idiopathic Parkinson's Disease, levodopa induced dyskinesia,; Levetiracetam, Keppra
MeSH Terms: conditions — Parkinson Disease | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
This is a 41-week trial composed of two consecutive parts (Part A, 14 weeks and optional Part B, 27 weeks) to evaluate the efficacy of levetiracetam in controlling levodopa induced dyskinesias in adults with Idiopathic Parkinson's Disease, without negative impact on the benefit on the motor function of the antiparkinsonian treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male / female adult, 30 years old or more;
2. Subject suffering from Idiopathic Parkinson's Disease, diagnosed according to the UK Brain Bank Criteria (see Appendix 14.8) (1) , since a minimum of 3 years, and stabilized with regard to the motor function (ratio .on./.off. over the day);
3. Subject treated with levodopa whether or not combined with any other antiparkinsonian drugs (except apomorphine) for minimum one year;
4. Subject experiencing during .on. periods, despite several attempts of treatment adjustment, persistent troublesome dyskinesias:

   1. with a minimum score of 2 on item 33 of the UPDRS-Part IV (moderately disabling dyskinesias);
   2. with a minimum score of 2 on item 32 of the UPDRS-Part IV (dyskinesias present during more than 25% of the waking day).

Exclusion Criteria:

1. Dyskinesias that cannot reliably be characterized on a regular basis by the subject himself/herself (more than 5 .errors. on DRC per 24 hours after repeated training);
2. Subject currently treated with apomorphine or neuroleptic drugs either typical or atypical such as clozapine, olanzapine or risperidone;
3. Subject currently treated with dopamine antagonists such as but not limited to metoclopramide, alizapride or phenothiazine derivatives (e.g. metopimazine). If necessary, the use of the dopamine antagonist domperidone is allowed.
4. Subject Who had undergone or who was scheduled for functional neurosurgery for Parkinson's disease during the trial period;

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of levetiracetam in controlling levodopa induced dyskinesias in adults with Idiopathic Parkinson's Disease by assessing the reduction in mean duration of dyskinesias during "on" period at 10-week

SECONDARY OUTCOMES:
Reduction in mean duration of dyskinesias per day at 9 month;Safety

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma